CLINICAL TRIAL: NCT05972564
Title: The Effect of SGLT2 Inhibition on Adipose Inflammation and Endothelial Function
Acronym: SADIE2
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Mona Mashayekhi, Assistant Professor, Division of Diabetes, Endocrinology and Metabolism, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 210907 (SADIE2)
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Metabolic Syndrome | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to placebo or empagliflozin in a 1:1 ratio, stratified for race and sex. A study biostatistician will prepare the randomization and allocation schedule.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo consists of gelatin capsules. To ensure blinding, empagliflozin will be over-encapsulated in identical gelatin capsules as placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin Arm (Active Comparator): Empagliflozin is an FDA-approved SGLT2 inhibitor used for the treatment of type 2 diabetes, with off-label use for diabetic kidney disease and for heart failure with reduced ejection fraction even in those without diabetes. To ensure blinding, empagliflozin will be over-encapsulated in identical gelatin capsules as placebo.
  Interventions: Drug: Empagliflozin 25 MG
- Placebo Arm (Placebo Comparator): Placebo consists of gelatin capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 25 MG — Empagliflozin is an FDA-approved SGLT2 inhibitor used for the treatment of type 2 diabetes, with off-label use for diabetic kidney disease and for heart failure with reduced ejection fraction even in those without diabetes.
  Other Names: Jardiance
  Arms: Empagliflozin Arm
Drug: Placebo — Placebo consists of gelatin capsules.
  Arms: Placebo Arm

SUMMARY:
Obesity is associated with increased cardiometabolic disease risk due, in part, to heightened chronic inflammation arising from adipose tissue. There are no current targeted therapies to prevent or reverse the chronic inflammation of obesity, and a better understanding of these inflammatory pathways in humans is key to future therapeutic interventions. This trial will determine both the anti-inflammatory potential of the SGLT2 inhibitor empagliflozin, and the contribution of adipose inflammation to surrogate measures of cardiovascular disease in a randomized controlled trial of obese patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years old
2. Metabolic syndrome as defined by 3 or more of 5 criteria:

   1. Systolic blood pressure ≥ 130 mmHg or diastolic blood pressure ≥ 85 mmg Hg or treatment with anti-hypertensive medications for minimum of 1 month
   2. Triglycerides ≥ 150 mg/dL or treatment with a triglyceride-targeted medication (fenofibrate, gemfibrozil, niacin, high dose omega-3 fatty acids)
   3. High-density lipoprotein (HDL) < 40 mg/dL in males or < 50 mg/dL in females
   4. Fasting blood glucose ≥ 100mg/dL or treatment with glucose-lowering medications
   5. Waist circumference ≥ 102 cm in males or ≥ 88cm in females
3. BMI ≥ 35 kg/M2
4. Scheduled gastric bypass or gastric sleeve in approximately 90 days (range 90-270 days)
5. The ability to provide informed consent

   Exclusion Criteria:
6. Type 1 diabetes.
7. Poorly controlled type 2 diabetes as defined by HbA1c ≥ 9%.
8. Use of anti-diabetic medications other than stable dose of metformin or a sulfonylurea in the last 1 month.
9. Treatment with a glucagon-like peptide-1 receptor agonist or co-agonist in the last 3 months.
10. Treatment with an SGLT2 inhibitor in the last 3 months.
11. Pregnancy or breast-feeding. Women of child-bearing potential will be required to have undergone surgical sterilization or to be using an intra-uterine device, hormonal contraceptive, or barrier methods of birth control.
12. Cardiovascular disease such as myocardial infarction within six months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (left ventricular hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, -second- or third-degree heart block, mitral valve stenosis, aortic stenosis, or hypertrophic cardiomyopathy
13. Presence of implanted cardiac defibrillator or pacemaker
14. History of serious neurologic disease such as cerebral hemorrhage, stroke, or transient ischemic attack
15. History of pancreatitis or pancreatic surgery
16. History or presence of immunological or hematological disorders
17. Clinically significant gastrointestinal impairment that could interfere with drug absorption
18. History of advanced liver disease with cirrhosis
19. Individuals with an eGFR<45 mL/min/1.73 m2, where eGFR is determined by the four-variable Modification of Diet in Renal Disease (MDRD) equation, where serum creatinine is expressed in mg/dL and age in years: eGFR (mL/min/1.73m2)=186 • Scr-1.154 • age-0.203 • (0.742 if female)
20. Treatment with chronic systemic glucocorticoid therapy (more than 7 consecutive days in 1 month)
21. Treatment with anticoagulants
22. Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult
23. History of alcohol abuse (>14 per week for men and >7 per week for women) or illicit drug use
24. Treatment with any investigational drug in the one month preceding the study
25. Previous randomization in this trial
26. Mental conditions rendering a subject unable to understand the nature, scope and possible consequences of the study
27. Inability to comply with the protocol in the opinion of the principal investigator, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

    Criteria Related to Known Adverse Effects of Drug:
28. Uncircumcised men or men with history of balanitis
29. History of urinary incontinence
30. History of recurrent (>3) episodes of vulvovaginitis per year, or severe symptoms
31. History of Fournier's gangrene
32. History of recurrent (≥3) UTIs per year or pyelonephritis
33. History of symptomatic hypotension or conditions predisposing to volume depletion
34. Known peripheral vascular disease, neuropathy, history of foot ulcers or lower limb amputations
35. Treatment with loop diuretics furosemide, torsemide, bumetanide, ethacrynic acid
36. Known or suspected allergy to trial medications, excipients, or related products
37. Contraindications to study medications, worded specifically as stated in the product's prescribing information

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Adipose tissue macrophages | 12 weeks
  Homeostatic adipose tissue macrophages are quantified
Flow mediated dilation | 12 weeks
  Brachial artery diameter is measured under basal conditions and during reactive hyperemia
Monocyte chemoattractant protein-1 | 12 weeks
  Plasma monocyte chemoattractant protein-1 levels are quantified

SECONDARY OUTCOMES:
Pro-inflammatory T cells | 12 weeks
  Pro-inflammatory T cells are quantified
IL-6 | 12 weeks
  Plasma IL-6 levels are quantified

CONTACTS AND LOCATIONS:
Overall Officials: Mona Mashayekhi, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD outside of VUMC study team.